CLINICAL TRIAL: NCT00900289
Title: DNA Methylation as a Predictor for Response and Progression-Free Survival in Patients With Ovarian Cancer
Brief Title: Studying DNA in Patients With Stage I, Stage II, Stage III, or Stage IV Ovarian Epithelial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liz-Anne Lewsley (Other)
Responsible Party: Sponsor-Investigator, Liz-Anne Lewsley, Project Manager, Cancer Research UK, Glasgow
Organization: Cancer Research UK, Glasgow (Other)
Other Study IDs: CDR0000577616; SCOTTISH-DNA-METHYLATION (Other: G75); EU-20793 (Other: EU)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cancer
Keywords: stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — DNA Methylation; Microarray Analysis; Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: microarray analysis
Genetic: polymerase chain reaction
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying tissue and blood samples from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This laboratory study is evaluating DNA to see how well it predicts response to treatment in patients with stage I, stage II, stage III, or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if DNA methylation patterns and expression of differentially methylated genes taken before chemotherapy can predict patient outcome with regard to progression-free survival.
* To evaluate whether DNA methylation can predict response assessed by RECIST criteria and CA 125 response.
* To evaluate the specificity and sensitivity of predicting methylation changes in tumor from the changes at the corresponding CpG islands in plasma.

OUTLINE: Tumor samples are collected at the time of initial laparotomy and blood is drawn prior to surgery for DNA methylation and biomarker studies.

Changes in DNA methylation will be examined globally using DNA methylation hybridization to microarrays and methylation specific PCR, as well as expression of genes shown to be differentially methylated.

ELIGIBILITY:
1. Clinically suspected FIGO stages Ic-IV epithelial ovarian cancer that are about to undergo surgery for confirmatory biopsy and attempted cytoreductive surgery
2. Given written informed consent
3. Female and >18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for this study will be patients with clinically suspected FIGO stages Ic-IV epithelial ovarian cancer that are about to undergo surgery for confirmatory biopsy and attempted cytoreductive surgery.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-03

PRIMARY OUTCOMES:
Progression-free survival | Ongoing
  To determine if DNA methylation patterns and expression differentially methylated genes taken before chemotherapy can predict patient outcome with regard to progression-free survival.

SECONDARY OUTCOMES:
Response | ongoing
  To evaluate whether DNA methylation can predict response.
Methylation changes in tumour | Ongoing
  To evaluate the specificity and sensitivity of predicting methylation changes in tumour from the changes at the corresponding CpG islands in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Siddiqui, MD, Principal Investigator — Scottish Gynaecological Cancer Trials Group
Locations (26):
- United Kingdom (26):
  - Basildon University Hospital, Basildon, England
  - St. Michael's Hospital, Bristol, England
  - Queens Hospital, Burton-on-Trent, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Derbyshire Royal Infirmary, Derby, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Hereford Hospitals, Hereford, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Barts and the London NHS Trust, London, England
  - Hammersmith Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - James Cook University Hospital, Middlesbrough, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Stirling Royal Infirmary, Stirling, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland